CLINICAL TRIAL: NCT04624347
Title: NEOVIDEO : Impact of Monitoring Motor Activity by Video Analysis on the Sleep of Very Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35RC18_8855_NEOVIDEO
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Infant Premature; Growth and Development; Neurologic Disorder; Sleep Fragmentation
MeSH Terms: conditions — Premature Birth; Nervous System Diseases; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Controlled, bicentric, single-blind, cross-over study with randomization of the sequence order (with and without caregivers' access to videos and movement curves).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acess to Videos and Movement curves (Experimental): with caregivers' access to videos and movement curves (4 days)
  Interventions: Behavioral: Access to video and movement curves
- No Acess to Video and Movement curves (No Intervention): without caregivers' access to videos and movement (4 days)

INTERVENTIONS:
Behavioral: Access to video and movement curves — intervention of caregivers with access to videos and motion curves of the premature infant
  Arms: Acess to Videos and Movement curves

SUMMARY:
Very premature birth and the necessary hospitalization expose to a risk of morbidity and mortality which impacts the neurodevelopmental prognosis. Sleep and behavior monitoring have not been developed in the neonatal units. This has to be improved since it is known from clinical and animal studies that the quality, organization and quantity of sleep in very preterm infants impact neurological development and brain plasticity.

The collection system provide neonatal care nurse with access to motion curves (evaluated by signal processing of live video) and real-time infrared video (also available in low-light conditions).

This new non-invasive technology allows an evaluation of the activity cycles of the newborn by the caregivers which until now was only accessible occasionally by short recordings of actigraphy or polysomnography. The investigators wish to demonstrate that this can contribute to an organization of care that respects the sleep patterns of the newborn, which they know to condition the neurodevelopmental prognosis.

DETAILED DESCRIPTION:
According to the EuroPeristat 2014 report, 1% of births are very preterm infants. Very premature birth and the necessary hospitalization expose to a risk of morbidity and mortality which impacts the neurodevelopmental prognosis. Sleep and behavior monitoring have not been developed in the neonatal units. This has to be improved since it is known from clinical and animal studies that the quality, organization and quantity of sleep in very preterm infants impact neurological development and brain plasticity. The publications suggest that alterations in sleep could have a significant impact on acquisitions in the areas of learning, memory, sensory development and behavior, as well as in the area of cardiorespiratory regulation. It has been shown that the implementation of developmental care practices (taking into account lighting, noise, the position of newborns and their rhythms) could have short-term beneficial effects on the sleep of very preterm infants. However, studies remain very limited in number. The investigators propose to build on the infrastructure developed as part of the H2020 DigiNewB project (http://www.digi-newb.eu/), which can provide neonatal care providers with access to motion curves (evaluated by signal processing of live video) and real-time infrared video (also available in low-light conditions).The collection system is functional, allows continuous analysis of videos to quantify movement and is suitable for incubators and neonatal beds. This new non-invasive technology allows an evaluation of the activity cycles of the newborn by the caregivers which until now was only accessible occasionally by short recordings of actigraphy or polysomnography. The investigators wish to demonstrate that this can contribute to an organization of care that respects the sleep patterns of the newborn, which they know to condition the neurodevelopmental prognosis.

ELIGIBILITY:
Inclusion Criteria:

New born :

* hospitalized in neonatology,
* at least one of whose legal representatives has given free, informed and written consent,
* term of birth <32 WA, postnatal age> 15 days and post-conceptual age between [30-38] WA,
* affiliated to a social security scheme

Caregivers:

* having at least 1 year of practical experience in neonatology,
* having been trained in the clinical basics of evaluating newborn sleep,
* having given their consent to participate.

Exclusion Criteria:

New born :

* sedative or curare treatment (opiates, benzodiazepines, curare, barbiturates) in the last 24 hours,
* chromosomal abnormalities identified
* Planned discharge date incompatible with the completion of the entire study

No criteria for caregivers

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Quantification of the percentage of time spent in sleep | for 8 days
  Quantification of the percentage of time spent in sleep (stage 1 + 2 of the neurobehavioral classification of Prechtl in 5 stages compared to the total duration of the analyzable tracing) by a supervised expert, viewing the blinded sequences of the condition tested (with and without access caregivers to video and movement curves).

SECONDARY OUTCOMES:
Quantification of the ratio of time spent in calm sleep / time spent in restless sleep . | for 8 days
  Prechtl stage 1 / stage 2 ratio
- Quantification of the percentage of time spent in the 5 stages of Prechtl / total analyzable tracing time. | for 8 days
- Quantification of sleep fragmentation and the different types of transitions: number and duration of awakening periods | for 8 days
- Quantification of sleep fragmentation and the different types of transitions: number and duration of movement periods (periods defined by successions of movements spaced less than 5 seconds apart) | for 8 days
  movement periods = periods defined by successions of movements spaced less than 5 seconds apart
- Quantification of sleep fragmentation and the different types of transitions: classification of all transitions between stages | for 8 days
- Care interventions: Quantification of the number and estimated stage of sleep at their initiation (in the 2 minutes preceding the intervention) | for 8 days
- Care interventions: Quantification of the duration and estimated stage of sleep at their initiation (in the 2 minutes preceding the intervention) | for 8 days
- Care interventions: Quantification of the type (noise or manual intervention) and estimated stage of sleep at their initiation (in the 2 minutes preceding the intervention) | for 8 days
- Textual analysis (lexical field) of the interview with the parents on their feelings about the device | At the end of 8 days recordings
- Textual analysis (lexical field) of the interview with the nursery nurses on their feelings about the device | At the end of 8 days recordings
- Analysis of the score of the "Ages and Stages questionnaires / Second Edition" sent to parents before their child's 24-month visit. | at 24 months
  Evaluate the child's skills in the various areas of his development. Questionnaire with 5 sections (Communication, Gross motor skills,Fine motor skills,Problem solving, Individual or social skills).
  Results sheet allowing rapid interpretation (positivity threshold for each sphere) and recommendations for each developmental area screened.

CONTACTS AND LOCATIONS:
Overall Officials: Céline CITTE, pediatric nurse, Principal Investigator — University Hospital of Rennes
Locations (2):
- France (2):
  - CHU Rennes Hôpital Sud, Rennes, Brittany Region
  - Pôle Femme Mère Enfant, Brest

IPD SHARING:
Plan to Share IPD: No